CLINICAL TRIAL: NCT04602884
Title: Early Detection of the 2019 Novel Coronavirus (SARS-CoV-2) Using Breath Analysis: First Cross-Sectional Study
Brief Title: Early Detection of COVID-19 Using Breath Analysis
Acronym: COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scentech Medical Technologies Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Cov-2-IDF
Record Dates: First submitted 2020-10-21; First posted 2020-10-26 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COVID-19 Positive patients (Experimental): subjects who were found COVID-19 Positive according to swab test.
  Interventions: Diagnostic Test: Breath biopsy sampling using the ReCIVA Breath Sampler
- Healthy subjects (Other): subjects who were found COVID-19 Negative according to swab test.
  Interventions: Diagnostic Test: Breath biopsy sampling using the ReCIVA Breath Sampler

INTERVENTIONS:
Diagnostic Test: Breath biopsy sampling using the ReCIVA Breath Sampler — Breath biopsy sampling using the ReCIVA Breath Sampler

SUMMARY:
EARLY DETECTION OF COVID-19 USING BREATH ANALYSIS- FIRST CROSS-SECTIONAL STUDY

DETAILED DESCRIPTION:
Primary objective- to identify and evaluate a set of biomarkers that represent both the genetic expression of the virus itself (SARS-CoV-2) and the metabolic activity of the immune system's response to the virus.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 55 years at the time of consent
* Positive results for SARS-CoV-2
* Capable of understanding written and/or spoken language
* Able to provide informed consent

Exclusion Criteria:

* Age under 18 years old
* (Anticipated) inability to complete breath sampling procedure due to e.g. hyper- or hypoventilation, respiratory failure, or claustrophobia when wearing the sampling mask
* Persons under guardianship or deprived of liberty
* Patients with the following diseases: Cancer, Asthma, Chronic Respiratory Disease
* Pregnant women
* Treated with antiviral drugs upon admission or during hospitalization
* Novices and soldiers in initial training

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Correlation between Volatile Organic Compounds pattern and COVID-19 detection status. | Through the study completion, up to 3 months.
  Correlation between the set of Volatile Organic Compounds found in breath biopsy and COVID-19 detection presence in a swab test.

SECONDARY OUTCOMES:
Correlation between Volatile Organic Compounds pattern and time from COVID-19 detection. | Through the study completion, up to 3 months.
  Correlation between the set of Volatile Organic Compounds found in breath biopsy and time since COVID-19 detected in a swab test.
Correlation between the set of Volatile Organic Compounds found in breath biopsy and disease intensity. | Through the study completion, up to 3 months.
  Correlation between the set of Volatile Organic Compounds found in breath biopsy and intensity of COVID-19 detected in a swab test.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Dror, PhD, Study Director — Scentech Medical Technologies Ltd
Locations (1):
- IDF COVID 19 Isolation Facility, Ashkelon, Israel

IPD SHARING:
Plan to Share IPD: No
No IPD is to be shared with other researchers.